CLINICAL TRIAL: NCT00755534
Title: A Parallel Phase II Study With Irinotecan/Cetuximab (Until PD) Followed by XELOX/Cetuximab (Until PD) vs the Reverse Sequence in Metastatic CRC With Previous Benefit on Irinotecan/Bevacizumab Based Therapy
Brief Title: Irinotecan/Cetuximab Followed by XELOX/Cetuximab vs the Reverse Sequence in Metastatic CRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.31
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer; Second line; Irinotecan; Cetuximab (Erbitux); Capecitabine (Xeloda)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Capecitabine; Cetuximab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Irinotecan+Erbitux -> XELOX+Erbitux
  Interventions: Drug: Irinotecan; Drug: Capecitabine; Drug: Cetuximab; Drug: Oxaliplatin
- 2 (Experimental): XELOX+Erbitux ->Irinotecan+Erbitux
  Interventions: Drug: Irinotecan; Drug: Capecitabine; Drug: Cetuximab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan (IV) 150 mg/m2 on day 1 every two weeks until progression
  Other Names: CPT-11; Campto
Drug: Capecitabine — Capecitabine (p.o) 2000 mg/m2 (1000 mg/m2 x 2) on day 1-7 every 2 weeks until progression
  Other Names: Xeloda
Drug: Cetuximab — Cetuximab(IV) 500 mg/m2 on day 1 every two weeks until progression
  Other Names: Erbitux
Drug: Oxaliplatin — Oxaliplatin (I.V) 85 mg/m2 on day 1 every two weeks until progression
  Other Names: Eloxatin; LoHP

SUMMARY:
This phase II study will evaluate which is the best way to administer cetuximab after recurrence in 1st line irinotecan+bevacizumab based treatment and to obtain results of the efficacy of the oxaliplatin+cetuximab combination as 2nd line treatment.

DETAILED DESCRIPTION:
Because of the recent advances in the field of systemic chemotherapy for mCRC, like irinotecan, oxaliplatin, capecitabine, and targeted agents (Cetuximab, Bevacizumab) mCRC patients have an overall survival that in some cases reaches 25 months.Irinotecan is an inhibitor of the DNA enzyme topoisomerase I, with use in clinical practice for the last 10 years.In a phase II study with mCRC patients resistant to irinotecan based therapy the combination of irinotecan and Cetuximab (an IgG1 anti-EGFR antibody) yielded a response rate of 22.5%.Capecitabine was shown to have improved tolerability and response rate compared with bolus 5-FU, with comparable time to progression and survival.Oxaliplatin has been approved by the FDA for 2nd line treatment in the metastatic CRC setting as a number of trials have shown promising data for response rates, disease stabilization rates,median progression free survival (PFS) and overall survival (OS).KRAS is a predictive marker for clinical benefit from EGFR-based antibody treatment. KRAS is the first molecular marker for selection of a targeted therapy in combination with a standard chemotherapy regimen. Patients with KRAS wild-type tumors have a strong benefit from the administration of cetuximab with better PFS and objective responses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal cancer
* Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* ECOG performance status ≤ 2
* Age 18 - 72 years
* Patients who have had a CR, PR or SD after 1st line therapy based on Irinotecan+Bevacizumab
* Paraffin block from the primary tumor in order to perform tha mutational analysis of the KRAS gene
* Adequate liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 4 upper normal limit, ALP ≤ 2.5 upper normal limit),renal (Creatinine ≤ 1.5 upper normal limit) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥100,000/mm3) function
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* Presence of central nervous system or brain metastases
* Pregnant or lactating woman
* Life expectancy < 3 months
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow or in the field where the treatment target is located
* Peripheral neuropathy grade ≥2
* Known hypersensitivity to Erbitux
* Metastatic infiltration of the liver >50%
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction or total colectomy
* Active infection
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Psychiatric illness or social situation that would preclude study compliance

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Time To Progression | 1 year

SECONDARY OUTCOMES:
Objective Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Toxicity profile | Toxicity assessment on each chemotherapy cycle
1 year Survival and Overall Survival | Probability of 1-year survival (%)
Correlation of the molecular characteristics of the tumor with the clinical outcome | Corralation after the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Heraklion, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - State General Hospital of Larissa, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki
  - Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki, Thessaloniki